CLINICAL TRIAL: NCT05134688
Title: Magnesium Sulphate for Tocolysis in Preterm Prelabour Rupture of Membranes
Brief Title: Magnesium Sulphate in Premature Rupture of Membranes
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Fathi Abdelraouf, Ahmed Fathi Abdelraouf, Assiut University
Other Study IDs: Magnesium sulphate in PPROM
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Premature Rupture of Membrane
Keywords: Magnesium sulphate
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grup 1: Group receive magnesium sulphate IV(4gm loading dose over 20 minutes followed by 1gm /hour for 6 hours
  Interventions: Drug: Magnesium sulfate
- Group 2: Receive no further treatment than conservative mangement( antibiotics and steroids)

INTERVENTIONS:
Drug: Magnesium sulfate — Tocolytic to stop preterm labor
  Groups: Grup 1

SUMMARY:
To assess the outcome of using magnesium sulphate on fetus and women with preterm premature rupture of membranes

DETAILED DESCRIPTION:
Preterm premature rupture of membranes (PPROM) is defined as rupture of the chorioamniotic membranes before the onset of labor prior to 37 weeks of gestation. Approximately 1% to 5% of pregnancies are complicated by PPROM . PPROM contributes to perinatal morbidity and mortality, secondary to premature birth, and maternal morbidity. Overall, PPROM accounts for about one-third of all preterm births . In order to reduce the effects of prematurity, early PPROM (24 to 33 weeks) is best served with conservative management in the absence of labor, infection, or fetal distress . The conservative management of PPROM consists of the use of antibiotic treatment and antenatal steroid to enhance fetal lung maturity . With or without the presence of labor, it is unclear whether tocolysis of women with PPROM would be efficacious in reducing the consequences of prematurity .The use of tocolytics in women with PPROM is still controversial. Many physicians use tocolytic therapy as a prophylactic measure and others initiate tocolysis only with the onset of contractions. There is also a variety of options for tocolysis: betamimetics, calcium channel blockers, cyclo-oxygenase (COX) inhibitors, oxytocin receptor antagonists and magnesium sulphate . As betamimetis is not available and isn't used in our country and magnesium sulphate is available magnesium sulphate is used widly. The loading dose of magnesium sulphate is IV 4 gm over 20 minutes followed by 1gm/hour for 6 hours The potential benefit from increased latency due to tocolysis must be weighed against the potential harm in increased maternal and perinatal infection, the latter of which can possibly lead to long-term sequelae for the child, including cerebral palsy

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with gastational age between 28 weeks and 36 weeks and 6 days who are diagnosed with preterm prelabour rupture of membranes

Exclusion Criteria:

* clinical suspicion of chorioamnionitis
* Patients refusal to participate in clinical research.
* significant vaginal bleeding
* previous tocolysis use after rupture of membranes
* nonreassuring fetal heart tracing
* fetal anomalies
* significant maternal medical complications, and maternal or fetal indication for delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Prospective cohort study
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Latency period after rupture of membranes | Baseline
  Measure letancy period between prelabour rupture of membranes and delivery during using magnesium sulphate as a tocolytic and without using magnesium sulphate

REFERENCES:
- [Background] Parry S, Strauss JF 3rd. Premature rupture of the fetal membranes. N Engl J Med. 1998 Mar 5;338(10):663-70. doi: 10.1056/NEJM199803053381006. No abstract available. PMID 9486996
- [Background] Kaltreider DF, Kohl S. Epidemiology of preterm delivery. Clin Obstet Gynecol. 1980 Mar;23(1):17-31. doi: 10.1097/00003081-198003000-00005. PMID 6988128
- [Background] ACOG Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 80: premature rupture of membranes. Clinical management guidelines for obstetrician-gynecologists. Obstet Gynecol. 2007 Apr;109(4):1007-19. doi: 10.1097/01.AOG.0000263888.69178.1f. PMID 17400872
- [Background] Crowther CA, Harding JE. Repeat doses of prenatal corticosteroids for women at risk of preterm birth for preventing neonatal respiratory disease. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003935. doi: 10.1002/14651858.CD003935.pub2. PMID 17636741
- [Background] McNamara HC, Crowther CA, Brown J. Different treatment regimens of magnesium sulphate for tocolysis in women in preterm labour. Cochrane Database Syst Rev. 2015 Dec 14;2015(12):CD011200. doi: 10.1002/14651858.CD011200.pub2. PMID 26662716
- [Background] Shatrov JG, Birch SCM, Lam LT, Quinlivan JA, McIntyre S, Mendz GL. Chorioamnionitis and cerebral palsy: a meta-analysis. Obstet Gynecol. 2010 Aug;116(2 Pt 1):387-392. doi: 10.1097/AOG.0b013e3181e90046. PMID 20664400
- [Background] Weiner CP, Renk K, Klugman M. The therapeutic efficacy and cost-effectiveness of aggressive tocolysis for premature labor associated with premature rupture of the membranes. Am J Obstet Gynecol. 1988 Jul;159(1):216-22. doi: 10.1016/0002-9378(88)90524-8. PMID 3134815